CLINICAL TRIAL: NCT04746885
Title: Effect of DHA on Proinflammatory Cytokines Including Platelets Activating Factor (PAF) and it's Role in Prevention of Necrotizing Enterocolitis in Preterm/Very Low Birth Weight Neonates
Brief Title: Effect of DHA on Proinflammatory Cytokines Including Platelets Activating Factor (PAF) in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DHA in preterm
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): (interventional group/ DHA): A minimum of 40 preterm infants will be included to receive 100mg DHA daily administered by enteral route for 30 days. This group will be subdivided into breast fed / artificially fed infants.
  Interventions: Dietary Supplement: DHA
- Group B (Other): (control group / Placebo): 40 of preterm infant controls will be included to receive placebo (physically matched solution). This group will be subdivided into breast fed / artificially fed infants.
  Interventions: Dietary Supplement: DHA

INTERVENTIONS:
Dietary Supplement: DHA — Oral supplement

SUMMARY:
The purpose of this study is to determine whether docosahexaenoic acid is effective in the prevention or reducing severity of necrotizing enterocolitis in preterm/low birth weight neonates.Necrotizing enterocolitis (NEC) is the most devastating gastrointestinal disease in neonates. The pathogenesis of NEC is not well defined but evidence strongly suggests that it is multifactorial . prematurity and enteral feeding are major risk factors for NEC. An excessive inflammatory response by the immature intestine to external stimuli, impaired intestinal barrier integrity and / or abnormal bacterial colonization are key factors implicated in pathophysiology of NEC.

DETAILED DESCRIPTION:
Inclusion criteria:

Patients are eligible for inclusion if they meet the following criteria:

Preterm neonates having a gestational age equal or less than 32 weeks at birth, admitted in Ain Shams University NICU'S.

Weight (less than or equal 1.500 KG) Clinically stable to begin enteral feeding All Genders (Male, Female) Written informed consent by parents Sepsis will not be considered as exclusion criteria (according to SNAP 11; this score considers six physiologic variables such as blood pressure, temperature, the Po2/Fio2 ratio, serum PH, seizures and urine output, Töllner score (table 3) and Rodwell score (table 4)).

Exclusion criteria:

Persistent bleeding at any level. Receiving medication to avoid coagulation. Persistent vomiting. Gastrointestinal malformations. Mother taking Omega-3 supplements and planning to breastfed. The enrolled patients will be subdivided into two groups; group A are infants receiving DHA, group B are infants receiving placebo (physically matched solution).

Our patient will be classified into two groups:

Group A (interventional group/ DHA):

A minimum of 40 preterm infants will be included to receive 100mg DHA daily administered by enteral route for 30 days. This group will be subdivided into breast fed / artificially fed infants.

Group B (control group / Placebo):

40 of preterm infant controls will be included to receive placebo (physically matched solution). This group will be subdivided into breast fed / artificially fed infants.

Sample size:

The sample size is calculated for the two groups receiving DHA versus Placebo. The sample size is calculated using the incidence densities of NEC reported in the literature of 4.4/1000 and 17.3/1000 baby day. At least 20 babies should be included in each arm to reach an effect size of 0.8 with alpha error = 0.05 and power 0.80 (G*Power 3.1.7, Franz Faul, Universität Kiel, Germany, 2013).

Randomization and blinding:

Group A and B assigned according to a predetermined schedule generated from random numbers based on a computer-generated randomization sequence into either DHA or Placebo.

Methods All infants will receive the standard neonatal care and will undergo follow-up from birth until reach 37 weeks corrected gestational age, discharge or death whichever comes first.

Feeding protocol: (Ellard and Anderson, 2012):

Begin as early as the neonate can tolerate.(when hemodynamically stable.) Start with low volume 0.5 to 1 ml/6 hours, increasing gradually according to the tolerance (trophic feeding 10-20 ml/kg) start deduction of feds from total fluid intake thereafter Gut priming is not used in patients with severe hemodynamic instability, suspected or confirmed NEC Increment from 10 to 20 ml/kg/day.

DHA supplementation:

Group (A): 100 mg DHA will be given to all neonates in group A as soon as possible with the enteral feeding for 30 days (subtracted from the total volume of the feed).

Group (B): will predominantly receive placebo (physically matched solution) together with their regular feeding.

All patients and controls subjected to:

Data Collection: Careful history taking Antenatal history including: rupture of membrane, Chorioamnionitis, history of urinary tract infection.

Natal history including: mode of delivery, place of delivery, the need for resuscitation, recorded Apgar score at 1minute and 5 minutes.

Postnatal history including: age of admission in neonatal intensive care unit, symptoms suggest infection.

Thorough clinical assessment:

Weight, length and OFC (twice weekly). Complete examination including cardiovascular, respiratory, and neurological examination.

Abdominal examination will done focusing on: signs of feeding intolerance including:

Measurement of abdominal girth Intestinal sounds Passage of stool Prescence of gastric residual Abdominal tenderness and rigidity NEC BELL'S criteria; as an objective tool for diagnosis and staging of NEC.

Laboratory investigations:

Complete blood picture, C-reactive protein, bleeding profile. Blood culture and sensitivity. Quantitative ELISA technique for PAF done for both cases and controls done twice. beseline sample will be withdrawn once NEC is suspected and the other one will be withdrawn 10 days from the first sample.( to assess the decrease in PAF levels).

BLOOD SAMPLES:

10ml of venous blood were withdrawn from each subject .they were divided into: 2ml collected on EDTA tube for CBC 1.8ml collected on sodium citrate for PT, PC and INR. The remaining part was collected in aplain tube, left to clot for 10-20 min at room temperature before centrifugation for 10 mins at the spend of 2000-3000 r.p.m., then serum was separated and divided into 2 aliquots, one for the blood chemistry which was assayed on the same day of sample collection, the second sample was stored at -20 C till the time of assay.

Radiological investigations:

Abdominal X-ray Erect & Supine (when necrotizing enterocolitis is suspected). Abdominal ultrasound (when necrotizing enterocolitis is suspected). MRI brain as an assessment tool for cerebral white matter abnormalities (White matter abnormalities scoring system).

Follow-up and end-point of the study:

1. Primary outcome:

   All infants will undergo follow-up from birth until reach 37 week corrected gestational age, discharge or death whichever comes first. The following primary outcome data will be recorded:

   Clinical examination and radiological investigations when clinically indicated for evidence of NEC.
2. A secondary outcome measure :

   Arthropemetric measures as weight increment per kg per week, length, OFC, duration of hospitalization, mortality if any, monitoring adverse effects of treatment (if any); such as emesis, increased gastric residuals, increased abdominal girth, diarrhea, skin rash. Long term outcome includes necrotizing enterocolitis, bronchopulmonary dysplasia and intracranial hemorrhage.

   At term equivalent, all preterm infants underwent a structural MRI scan that was analysed qualitatively for the prescence and severity of cerebral white matter abnormalities, including cysts, signal abnormalities, loss of white matter volume, ventriculomegally, and corpus callosal thinning/myelination. (Each infant's scan was then graded using a qualitative scoring system consisting of five 3-point scales assessing the presence and severity of periventricular white matter volume loss, white matter signal abnormality, the presence of cystic abnormalities, ventricular dilation, and thinning of the corpus callosum and reduced myelination . children were classified as follows: 1) no abnormalities (score of 5 to 6) ; 2) mild abnormalities (score of 7 to 9) ; 3) moderate abnormalities (score of 10 to12) ; or 4) severe abnormalities (score >12).
3. Tertiary outcome:

After discharge, all children underwent a comprehensive neurodevelopmental assessment using Bayley scale of infant and Toddler Development -111 (Bayley-111)

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates having a gestational age equal or less than 32 weeks at birth, admitted in Ain Shams University NICU'S.

Weight (less than or equal 1.500 KG) Clinically stable to begin enteral feeding All Genders (Male, Female) Written informed consent by parents Sepsis will not be considered as exclusion criteria (according to SNAP 11; this score considers six physiologic variables such as blood pressure, temperature, the Po2/Fio2 ratio, serum PH, seizures and urine output, Töllner score (table 3) and Rodwell score

Exclusion Criteria:

* Persistent bleeding at any level. Receiving medication to avoid coagulation. Persistent vomiting. Gastrointestinal malformations. Mother taking Omega-3 supplements and planning to breastfed.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
DEVELOPMENT OF NEC | 3-10 DAYS
  All infants will undergo follow-up from birth until reach 37 week corrected gestational age, discharge or death whichever comes first. The following primary outcome data will be recorded:
  Clinical examination and radiological investigations when clinically indicated for evidence of NEC.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Aderem A, Ulevitch RJ. Toll-like receptors in the induction of the innate immune response. Nature. 2000 Aug 17;406(6797):782-7. doi: 10.1038/35021228. PMID 10963608
- [Result] Meguro A, Kuribayashi R, Sakurada T, Sekine T, Aida H, Abe T. [Intravascular hemolysis due to residual shunt after patch closure of VSD: a case report]. Kyobu Geka. 1992 Jun;45(6):537-40. Japanese. PMID 1602686
- [Result] Axelsson A, Lindgren F. [Firecrackers--a risk of hearing injuries?]. Lakartidningen. 1987 Apr 15;84(16):1341-6. No abstract available. Swedish. PMID 3586783
- [Result] Miles EA, Calder PC. Modulation of immune function by dietary fatty acids. Proc Nutr Soc. 1998 May;57(2):277-92. doi: 10.1079/pns19980042. No abstract available. PMID 9656331